CLINICAL TRIAL: NCT00461214
Title: General Surgery Training Outcomes Project: Evaluating the Impact of the Curriculum on General Surgery Resident Training and Evaluation
Brief Title: General Surgery Training Outcomes Project
Status: Terminated | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Dennis Fowler, Professor of Clinical Surgery, Columbia University
Other Study IDs: AAAC1896
Record Dates: First submitted 2007-04-13; First posted 2007-04-17 (Estimated); Last update posted 2012-11-21 (Estimated); Status verified 2012-11

CONDITIONS: Healthy
Keywords: laparoscopy; surgery; technical skills; outcomes; resident training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Participation in laparoscopic training curriculum — General Surgery Training Outcome

SUMMARY:
The purpose of the General Surgery Training Outcomes Project: Evaluating the Impact of the Curriculum on General Surgery Resident Training and Evaluation is to analyze data collected as a normal course of the general surgery curriculum. The information collected is data readily available and routinely collected on all participants in the general surgery curriculum at NewYork Presbyterian Hospital/Columbia Campus. This information may lead to improvement in the general surgery curriculum.

ELIGIBILITY:
Inclusion Criteria:

* All general surgery interns and PGY2-5's at NewYork Hospital/Columbia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgery interns and PGY2-5's
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2006-10; Primary Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis L Fowler, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University College of Physicians and Surgeons, New York, New York, United States